CLINICAL TRIAL: NCT05838053
Title: Comparison of Segmentectomy Versus Lobectomy for Lung Adenocarcinoma ≤ 2cm With Micropapillary and Solid Subtype Positive by Frozen Section: A Prospective, Observational, Multicenter Cohort Study
Brief Title: Comparison of Segmentectomy Versus Lobectomy for Lung Adenocarcinoma ≤ 2cm
Status: Recruiting | Type: Observational
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Deping Zhao, Director of thoracic surgery; Principal Investigator, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: STAR 002
Record Dates: First submitted 2023-04-20; First posted 2023-05-01 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Lung Adenocarcinoma
Keywords: frozen sections; lobectomy; segmentectomy; micropapillary
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — Mastectomy, Segmental

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lobectomy with systemic lymph node dissection: lobectomy with hilar and mediastinal lymph node dissection is performed. Systemic or selective lymph node dissection is mandatory, and nodal sampling is not allowed. At least three stations of mediastinal lymph node from 2R, 4R, 7, 8, 9 for the right side and 5, 6, 7, 8, 9 for the left side, respectively.
  Interventions: Procedure: Lobectomy with systemic lymph node dissection
- Segmentectomy with systemic lymph node dissection: Segmentectomy with hilar and mediastinal lymph node dissection is performed. If the tumor located at inter-segment plane and without sufficient resection margin distance, a combined segmentectomy will be performed after a comprehensive evaluation. As with lobectomy, systemic or selective lymph node dissection is mandatory, and nodal sampling is not allowed. At least three stations of mediastinal lymph node from 2R, 4R, 7, 8, 9 for the right side and 5, 6, 7, 8, 9 for the left side, respectively. The distance from the dissection margin to the tumor edge must be evaluated in the same manner as with lobectomy.
  Interventions: Procedure: Segmentectomy with systemic lymph node dissection

INTERVENTIONS:
Procedure: Lobectomy with systemic lymph node dissection — Lobectomy with hilar and mediastinal lymph node dissection is performed. Segmentectomy with hilar and mediastinal lymph node dissection is performed. Systemic or selective lymph node dissection is mandatory, and nodal sampling is not allowed. At least three stations of mediastinal lymph node from 2R, 4R, 7, 8, 9 for the right side and 5, 6, 7, 8, 9 for the left side, respectively. The distance from the dissection margin to the tumor edge must be evaluated intra-operatively. If the distance is either less than the maximum tumor diameter or 20 mm, the absence of cancer cells in the resection margin must be histologically or cytologically confirmed before finishing surgery.
  Groups: Lobectomy with systemic lymph node dissection
Procedure: Segmentectomy with systemic lymph node dissection — Segmentectomy with hilar and mediastinal lymph node dissection is performed. If the tumor located at inter-segment plane and without sufficient resection margin distance, a combined segmentectomy will be performed. Systemic or selective lymph node dissection is mandatory, and nodal sampling is not allowed. At least three stations of mediastinal lymph node from 2R, 4R, 7, 8, 9 for the right side and 5, 6, 7, 8, 9 for the left side, respectively. The distance from the dissection margin to the tumor edge must be evaluated intra-operatively. If the distance is either less than the maximum tumor diameter or 20 mm, the absence of cancer cells in the resection margin must be histologically or cytologically confirmed before finishing surgery.
  Groups: Segmentectomy with systemic lymph node dissection

SUMMARY:
This study aims to evaluate the superiority in recurrence-free survival of lobectomy compared with segmentectomy in patients with lung adenocarcinoma ≤ 2 cm with micropapillary and solid subtype positive by intraoperative frozen sections.

DETAILED DESCRIPTION:
At present, the technology of intraoperative frozen section has gradually matured, which can diagnose the benign and malignant tumors and guide the resection strategy for peripheral small-sized lung adenocarcinoma. Travis et al. reported high specificity of intraoperative frozen section in the identification of micropapillary components, confirming that intraoperative frozen section may guide the selection of surgical procedures. However, there is still little evidence whether segmentectomy is appropriate for invasive adenocarcinoma without micropapillary patterns. This prospective and multi-center study was aimed to evaluate the superiority in recurrence free survival and overall survival of lobectomy compared with segmentectomy in patients with lung adenocarcinoma (≤ 2 cm) containing positive micropapillary components.

ELIGIBILITY:
Inclusion Criteria:

* Tumor size ≤ 2 cm;
* Solitary tumor and located in the outer third of the lung field;
* Preoperative CT indicated that the nodules were single nodules or Concomitant nodules was less than minimal invasive adenocarcinoma;
* Intraoperative frozen section confirmed invasive lung adenocarcinoma and with micropapillary and solid patterns positive (>5%);
* Confirmation of R0 status by intraoperative frozen section analysis;
* Pulmonary function could withstand both segmentectomy and lobectomy (FEV1 > 1.5 L or FEV1% ≥ 60%);
* Sufficient organ function;
* Performance status of 0,1 or 2；
* Written informed consent.

Exclusion Criteria:

* The tumor is close to the hilum, which cannot perform segmentectomy ;
* Patients suspected of lymph node positive by preoperative examination, including CT scans and mediastinal lymph node biopsy;
* Evidence revealed locally advanced or metastatic disease;
* Intraoperative exploration revealed accidental pleural dissemination.
* Patients with severe damage to heart, liver and kidney function (grade 3 ~ 4, Alanine aminotransferase (ALT) and/or Aspartate aminotransferase (AST) over 3 times the normal upper limit, Cr over the normal upper limit).
* Patients concomitant with other malignant tumors；
* Patients had prior chemotherapy, radiotherapy or molecular targeted therapy for this malignancy.
* History of severe heart disease, heart failure, myocardial infarction within the past 6 months.
* The patients who were not suitable for inclusion by researchers' evaluation.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: clinical stage IA patients with Lung Adenocarcinoma ≤ 2cm as well as micropapillary and solid Subtype positive (>5%) by frozen sections
Sampling Method: Non-Probability Sample
Enrollment: 446 (Estimated)
Dates: Start 2019-08-20 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
recurrence-free survival rate | 5 year
  Recurrence-free survival (RFS) was defined as the time from surgery until recurrence or death from any cause

SECONDARY OUTCOMES:
overall survival rate | 5 year
  Overall survival (OS) was defined as the time from surgery until death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Yangpu, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided